CLINICAL TRIAL: NCT02907801
Title: Effects of Perception-Action Approach Intervention in Infants With Congenital Muscular Torticollis: A Randomized Nonconcurrent Multiple Baseline Study
Brief Title: Perception-Action Approach Intervention for Infants With Congenital Muscular Torticollis
Acronym: P-AA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: After a reliability pilot, main study stopped due to unrelated clinic closure.
Sponsor: Rosalind Franklin University of Medicine and Science (Other)
Collaborators: Ability Pediatric Physical Therapy, LLC (Other)
Responsible Party: Principal Investigator, Mary Rahlin, Associate Professor, Rosalind Franklin University of Medicine and Science
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 433 PT
Record Dates: First submitted 2016-09-13; First posted 2016-09-20 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Congenital Muscular Torticollis
Keywords: congenital muscular torticollis; infants; perception-action approach
MeSH Terms: conditions — Congenital torticollis | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Perception-Action Approach (Experimental): Perception-Action Approach (P-AA) intervention components include environmental set-up for activity and participation in play, manual guidance in the form of light pressure applied to the infant's body in developmentally appropriate positions, and caregiver education in modifications to everyday activities consistent with the P-AA. All components are designed to promote spontaneous exploration of the environment by the infant by suggesting small, incremental changes in his/her perceptual-motor orientation and contact with the support surface. Intervention is progressed by gradually removing the environmental supports and therapist's hands to allow for spontaneous exploration of a newly found contact with the support surface or new body configuration.
  Interventions: Behavioral: Perception-Action Approach

INTERVENTIONS:
Behavioral: Perception-Action Approach — Environmental set-up, gentle manual guidance, and caregiver education
  Other Names: Perceptual-motor intervention, physical therapy

SUMMARY:
Infants with congenital muscular torticollis (CMT) display postural and functional asymmetry that interferes with their development. The use of the Perception-Action Approach (P-AA) intervention in infants with CMT is supported by a single case report and needs to be researched further to determine its efficacy. This study will investigate the immediate effects of the P-AA intervention on habitual head deviation from midline, active head rotation range of motion, and functional use of both sides of the body in infants with CMT.

The participants will be 3 infants with CMT, aged birth to 9 months. A randomized, nonconcurrent A-B multiple baseline design across subjects will be used. The intervention phase will include 5 daily PT sessions, with outcome data collected at the end of each session.

It is hypothesized that improvements on all outcome measures will be documented upon the initiation of the P-A Approach intervention, with the most substantial change expected in habitual head deviation from midline measured by still photography.

DETAILED DESCRIPTION:
This study will have a randomized, nonconcurrent A-B multiple baseline design across subjects. The purpose of this study will be to investigate the immediate effects of the P-AA intervention on habitual head deviation from midline, active head rotation range of motion (ROM), and functional use of both sides of the body in infants with CMT.

The participants will be 3 infants with CMT, aged birth to 9 months, recruited from a private pediatric physical therapy (PT) practice. Baseline and intervention data will be collected 5 days per week, Monday through Friday, until the study is completed. The length of the baseline phase will be randomly assigned to each consecutively enrolled participant. The appropriate measurements will be taken at every baseline phase session but no intervention will be provided until the intervention phase is initiated. The intervention phase will include 5 daily PT sessions during which the P-AA intervention will be used, with outcome data collected at the end of each session. Additionally, the participants' therapy-related behavior during intervention sessions will be documented.

Measurements of still photos and scoring of video recordings to evaluate the participants' habitual head deviation from midline and functional use of both sides of the body for movement and play will be performed by an assessor blind to the timing of when the photos and videos are obtained within the study. The active head rotation ROM measurements and assessment of therapy-related behavior will be performed by the treating therapists.

Prior to initiating this research, a pilot reliability study will be conducted for all outcome measures. A total of 3 to 5 infants will be recruited for the pilot project.

Fidelity of intervention will be evaluated during the pilot study using a checklist. During the main study, intervention adherence will be assessed by tracking attendance, session duration, and intervention frequency.

ELIGIBILITY:
Inclusion Criteria:

* age between birth and 9 months at the time of recruitment
* diagnosis of CMT as documented in the medical record
* parents/guardians agree not to have their child participate in any additional interventions for CMT during the course of the study

Exclusion Criteria:

* diagnosis of neuromuscular torticollis, Sandifer syndrome, acute torticollis, benign paroxysmal torticollis, ocular torticollis, torticollis related to bony anomalies, or another non-muscular type of torticollis
* being seen for torticollis by another health care provider
* receiving a passive stretching intervention for CMT prior to referral for PT at the research site

Max Age: 9 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2017-01-10 (Actual); Primary Completion 2018-03-26 (Actual); Study Completion 2018-03-26 (Actual)

PRIMARY OUTCOMES:
Still Photography | Up to 12 days (assessed at every baseline session and at the end of every intervention session for a total of 10, 11 or 12 sessions, depending on the length of the baseline phase)
  Change in the angle of habitual head deviation from midline assessed in a supine position
Arthrodial Goniometry | Up to 12 days (assessed at every baseline session and at the end of every intervention session for a total of 10, 11 or 12 sessions, depending on the length of the baseline phase)
  Change in the angular difference in active cervical rotation range of motion between the involved and uninvolved sides
Functional Symmetry Observation Scale (FSOS) | Up to 12 days (assessed at every baseline session and at the end of every intervention session for a total of 10, 11 or 12 sessions, depending on the length of the baseline phase)
  Change in the FSOS score that reflects functional use of both sides of the body during spontaneous movement and play

SECONDARY OUTCOMES:
Therapy Behavior Scale (TBS), Version 2.2 | 5 days (assessed after each of 5 intervention sessions)
  The TBS score documents therapy-related behavior during intervention sessions

CONTACTS AND LOCATIONS:
Overall Officials: Mary Rahlin, PT, DHS, PCS, Principal Investigator — Rosalind Franklin University of Medicine and Science
Locations (1):
- Ability Pediatric Physical Therapy, LLC, Anchorage, Alaska, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kaplan SL, Coulter C, Fetters L. Physical therapy management of congenital muscular torticollis: an evidence-based clinical practice guideline: from the Section on Pediatrics of the American Physical Therapy Association. Pediatr Phys Ther. 2013 Winter;25(4):348-94. doi: 10.1097/PEP.0b013e3182a778d2. PMID 24076627
- [Background] Rahlin M. TAMO therapy as a major component of physical therapy intervention for an infant with congenital muscular torticollis: a case report. Pediatr Phys Ther. 2005 Fall;17(3):209-18. doi: 10.1097/01.pep.0000179176.20035.f0. PMID 16357675
- [Background] Tscharnuter I. Clinical Application of Dynamic Theory Concepts According to Tscharnuter Akademie for Movement Organization (TAMO) Therapy. Pediatr Phys Ther. 2002 Spring;14(1):29-37. PMID 17053679
- [Background] Romeiser Logan L, Hickman RR, Harris SR, Heriza CB. Single-subject research design: recommendations for levels of evidence and quality rating. Dev Med Child Neurol. 2008 Feb;50(2):99-103. doi: 10.1111/j.1469-8749.2007.02005.x. PMID 18201299
- [Background] Rahlin M, Sarmiento B. Reliability of still photography measuring habitual head deviation from midline in infants with congenital muscular torticollis. Pediatr Phys Ther. 2010 Winter;22(4):399-406. doi: 10.1097/PEP.0b013e3181f9d72d. PMID 21068640
- [Background] Rahlin M, McCloy C, Henderson R, Long T, Rheault W. Development and content validity of the Therapy Behavior Scale. Infant Behav Dev. 2012 Jun;35(3):452-65. doi: 10.1016/j.infbeh.2012.03.001. Epub 2012 Jun 26. PMID 22729134